CLINICAL TRIAL: NCT03685032
Title: Effects of Intraoperative Dexamethasone and Ondansetron on Postoperative Nausea and Vomiting in Microvascular Decompression Surgery: A Randomized Controlled Study
Brief Title: Effects of Intraoperative Dexamethasone and Ondansetron on Postoperative Nausea and Vomiting in Microvascular Decompression Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Clinical Assistant Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE571218
Record Dates: First submitted 2018-09-23; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Microvascular Decompression Surgery; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Ondansetron; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized control trial was conducted. The investigators allocated patients into two arm.
  The study group (Gr. D) received intraoperative dexamethasone 4 mg iv and ondansetron 4 mg iv, whereas the control group (Gr. N) received placebo (0.9% normal saline 1 ml iv and 0.9% normal saline 2 ml iv)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study drugs based on a sequentially numbered list were prepared in the same way. These drugs had similar characteristics, including clear color and no observable particles, and were loaded into syringes labeled for each group. The attending anesthesiologists, anesthetic nurses, and ward nurses, as well as the patients were blinded to the computer-generated randomization lists.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Gr. D) (Experimental): After patients received general anesthesia, a sequentially numbered opaque sealed envelope was opened. Gr. D was administered 4 mg of dexamethasone in 1 ml iv.
  At the end of the operation when suturing the dura mater, Gr. D received ondansetron 4 mg in 2 ml iv.
  Interventions: Drug: Dexamethasone; Drug: Ondansetron
- the control group (Gr. N) (Placebo Comparator): After patients received general anesthesia, a sequentially numbered opaque sealed envelope was opened. Gr. N received normal saline 1 ml iv.
  At the end of the operation when suturing the dura mater, Gr. N received normal saline 2 ml iv.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Dexamethasone — The 4 mg of dexamethasone in 1 ml intravenous was administrated after patient received general anesthesia
  Other Names: Lodexa
  Arms: The study group (Gr. D)
Drug: Ondansetron — The 4 mg of ondansetron in 2 ml intravenous was administrated at the end of the operation.
  Other Names: Onsia
  Arms: The study group (Gr. D)
Drug: 0.9% Sodium Chloride Injection — The 0.9% sodium chloride in 1 ml intravenous was administrated after patient received general anesthesia. At the end of operation, the 0.9% sodium chloride in 2 ml intravenous was administrated.
  Arms: the control group (Gr. N)

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common problem and may lead to catastrophic complications, especially in neurosurgical cases. The aim of this study was to evaluate the effects of dexamethasone and ondansetron for preventing PONV in patients who underwent microvascular decompression surgery (MVD).

DETAILED DESCRIPTION:
A prospective, double-blinded randomized control trial was conducted with 54 patients who underwent MVD. Patients were allocated into two groups. The study group (Gr. D) received intraoperative dexamethasone 4 mg iv and ondansetron 4 mg iv, whereas the control group (Gr. N) received placebo (0.9% normal saline 1 ml iv and 0.9% normal saline 2 ml iv). The incidence and severity of PONV were observed at 1, 2, 4 and 24 hr post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for MVD of trigeminal nerve root
* Patients who had a physical status classification of I to III according to the American Society of Anesthesiologists, and those who had a body mass index of 18 to 35 kg/m2

Exclusion Criteria:

* Patients on long-term administration of dexamethasone or ondansetron, those with a history of allergic reactions to dexamethasone or ondansetron, those who had undergone antiemetic therapy within 24 hr before surgery, those with underlying liver or renal failure, those who were pregnant, or those who had undergone emergency surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-08-07 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2016-02-16 (Actual)

PRIMARY OUTCOMES:
Change in incidence of postoperative nausea and vomiting | The incidence was recorded at 1 hour as a baseline and changing incidences from baseline were recorded at 2 hours, 4 hours, and 24 hours.
  Postoperative nausea and vomiting events was recorded by blinded anesthesiologists, blinded anesthetic nurses, and blinded ward nurses.

SECONDARY OUTCOMES:
Pain score | The intensity of pain was recorded at 1 hour and 2 hours in the postoperative period in the recovery room and at 4 hours and 24 hours in the ward.
  The intensity of postoperative pain was measured with a numeric rating scale (NRS: 0=no pain, 10=severe pain)
opioid analgesics consumed | The opioid analgesics used was recorded at 1 hour and 2 hours in the postoperative period in the recovery room and at 4 hours and 24 hours in the ward.
  opioid analgesics consumed was recorded by blinded anesthesiologists, blinded anesthetic nurses, and blinded ward nurses.
severity of postoperative nausea and vomiting | The severity of postoperative nausea and vomiting was recorded at 1 hour and 2 hours in the postoperative period in the recovery room and at 4 hours and 24 hours in the ward.
  Severity of postoperative nausea and vomiting was recorded by blinded anesthesiologists, blinded anesthetic nurses, and blinded ward nurses. Level of severity of PONV (0=no symptoms; 1=mild: few symptoms and not requiring treatment; 2=moderate: presented symptoms and needed ondansetron 8 mg iv; 3=severe: persisted symptoms after received ondansetron 8 mg iv and needed re-administration of ondansetron 8 mg iv)
Antiemetics used | The antiemetic used was recorded at 1 hour and 2 hours in the postoperative period in the recovery room and at 4 hours and 24 hours in the ward.
  Antiemetics used was recorded by blinded anesthesiologists, blinded anesthetic nurses, and blinded ward nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Pornthep Kasemsiri, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

REFERENCES:
- [Background] Ha SH, Kim H, Ju HM, Nam DJ, Min KT. Comparison of the antiemetic effect of ramosetron with ondansetron in patients undergoing microvascular decompression with retromastoid craniotomy: a preliminary report. Korean J Anesthesiol. 2015 Aug;68(4):386-91. doi: 10.4097/kjae.2015.68.4.386. Epub 2015 Jul 28. PMID 26257852